## Are Sugar-Sweetened Beverage Information Labels Well-Targeted? NCT05038163

Informed Consent Form
August 17<sup>th</sup>, 2021

## **Informed Consent Form**

Thanks for your interest! This is a research study by Dmitry Taubinsky from the University of California. We're interested to know what kinds of drinks people like, as part of a study on consumer choice patterns. If you agree to participate, we'll ask you some background questions and ask you to choose between different drinks.

You must take this survey on a tablet, laptop, or desktop computer, not on a mobile phone.

This survey has two parts. If you participate, you'll take Part 1 now, and we will email you a link to take Part 2 in a few days. Each part takes about 10 minutes.

Please do not try to take this survey more than once. We have ways to detect this, and we will not pay people for taking the survey again.

After you complete Part 2, we will pay you \$15 using an online gift card and possibly a 12-pack of drinks. Specifically, one third of respondents will be randomly selected to receive a 12-pack of drinks they chose in one of the survey questions plus an online gift card for the difference between \$15 and the price of the drinks. The remaining respondents will receive their entire \$15 reward in the form of an online gift card. For those who are selected to receive drinks, we will send the drinks to your address directly from either Walmart or Amazon. Thus, you should only participate in this study if you are interested in receiving drinks after the study is over.

You will only be paid if you complete both surveys and answer correctly on the "attention check" question(s).

This study will be registered at ClinicalTrials.gov within 21 days of the first subject's enrollment. We will post the anonymized data from this study at ClinicalTrials.gov and, potentially, in other research data repositories. Before posting the data, we will remove any information that could identify you personally.

Participation in this study is completely voluntary. You are free to decline to participate or to end participation at any time for any reason. If you have questions, comments, or complaints about this study, feel free to contact Daniel Cohen at daniel.m.cohen@berkeley.edu. The identifying number for this survey is CPHS# 2020-08-13558.

Are you willing to participate in this survey?

- Yes, I am willing to participate.
- No, I am not willing to participate.